CLINICAL TRIAL: NCT06693193
Title: Personalized Virtual Environments for Patients with Cognitive Impairment Exhibiting Responsive Behaviors: Proof-of-Concept and Feasibility Study
Brief Title: Personalized Virtual Environments for Managing Responsive Behaviors in Cognitively Impaired Patients: a Feasibility Study
Acronym: iEMBRACE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Bruno Kessler (Other)
Responsible Party: Principal Investigator, Susanna Pardini, Researcher, Fondazione Bruno Kessler
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: VR2024
Record Dates: First submitted 2024-11-12; First posted 2024-11-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Cognitive Impairment; Dementia
Keywords: Customization; Customized Virtual Reality Scenarios; Cognitive Impairment; Responsive Behaviors; Virtual Reality Therapy; Non pharmacological therapy
MeSH Terms: conditions — Cognitive Dysfunction; Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (1):
- Virtual Reality group (Experimental): Participants will undergo three VR exposure sessions using Oculus headsets, presenting a virtual environment with realistic natural stimuli or customized environments tailored to individual preferences and valued activities. For each environment, auditory (e.g., animal sounds, wind rustling, type of music) and visual elements (e.g., presence of people, objects, or animals), as well as time of day and weather conditions, can be adjusted. The operator will customize the environment through a user-friendly smartphone app interface, enabling real-time parameter adjustments and content selection. During VR exposure, the operator can observe the participant's visual focus in real-time.
  Interventions: Device: Immersive Virtual Reality

INTERVENTIONS:
Device: Immersive Virtual Reality — Individuals will participate in three VR sessions using Oculus headsets, experiencing virtual environments featuring realistic natural stimuli or custom settings tailored to their preferences and valued activities. Each environment allows for the adjustment of auditory elements (such as animal sounds, rustling wind, or specific music), visual elements (such as people, objects, or animals), and the time of day and weather conditions. The operator will use a user-friendly smartphone app to customize the environment, making real-time adjustments to settings and content. Throughout the VR experience, the operator can monitor the participant's visual focus in real-time.

SUMMARY:
The goal of this feasibility study is to explore the feasibility of using realistic, customizable virtual reality (VR) environments in response to the onset of Responsive Behaviors in elderly residents with cognitive impairment.

Specifically, the study will assess;

* feasibility through acceptance metrics (including recruitment rate, adherence rate, attrition rate, and tolerance to the intervention);
* safety (monitoring for adverse effects related to VR headset use);
* user engagement, enjoyment, and overall experience.

Participants will be exposed to three VR sessions conducted before, during, or after a situation deemed activating (e.g., personal hygiene activities). Operators will conduct a baseline assessment to identify specific moments when the participant experiences responsive behaviors. Additionally, operators may administer the Oculus VR headset when responsive behaviors occur outside of baseline-identified moments.

DETAILED DESCRIPTION:
Study Site and Environment: Data collection will occur at the Azienda Pubblica di Servizi alla Persona "Margherita Grazioli" in Povo, Trento. The experimental setup will be free from external interference to minimize distractions and ensure a smooth study process. The study will be conducted in familiar, ecologically relevant settings within APSP, selecting environments likely to stimulate activation states in participants.

Duration and Procedure: The study is expected to last six months. Each participant will undergo at least three VR sessions about situations that may trigger activation, such as personal hygiene activities. A baseline assessment will pinpoint specific times when participants exhibit responsive behaviors. Additionally, VR sessions may be initiated if responsive behaviors arise outside the predicted times using the Oculus headset.

Procedure and Timing for Each VR Session:

Preliminary Assessment (Participant Selection) (~30 minutes):

Participants are selected based on inclusion/exclusion criteria and provided with informed consent.

Information is collected from clinical records and updated based on the participant's condition.

An initial assessment examines responsive behaviors' type, frequency, and timing using demographic information, FAST, NPI, and CMAI.

Pre-Session Evaluation (T0) (~15 minutes):

Assessments include pain, responsive behaviors, emotions, anxiety, pleasantness, and discomfort before VR use (using PAINAD and STAI-Y1).

Virtual Environment Selection (~5 minutes):

The operator selects the VR environment for the participant through a smartphone linked to the Oculus headset via WiFi.

Procedure Explanation and Contextualization (~5 minutes):

A brief overview of the session and VR setup is provided to the participant.

Familiarization with Oculus Headset (~1-2 minutes):

A brief period to help the participant acclimate to the VR headset.

VR Session and During-Session Evaluation (T1) (~8 minutes within tolerance):

The VR session is audio-visual recorded, with the operator noting participant behaviors and responses (using OERS, Observation Sheet, STAI-Y1, Ad Hoc Questionnaire, PAINAD, and DataSheet2).

Post-Session Evaluation (T2) (~15 minutes):

Pain, responsive behaviors, emotions, anxiety, pleasantness, and discomfort are re-evaluated (using PAINAD, DataSheet2, Ad Hoc Questionnaire, STAI-Y1, OERS, NPT-ES, and VRSQ).

Final Evaluation (T3) (~10 minutes):

After all sessions, a final assessment using the Cohen-Mansfield Agitation Inventory (CMAI) is conducted.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18 years of age.
* Native Italian speakers.
* Can provide written informed consent for study participation or have a legal guardian who can give consent on their behalf.

Exclusion Criteria:

* Presence of any psychiatric diagnoses as recorded in medical records.
* A total score of ≥ 40 on the Neuropsychiatric Inventory (NPI) indicates neuropsychiatric symptoms.
* A partial NPI score > 6 in the domains of agitation/aggression or delusions.
* Enrollment in palliative care services.
* Severe neurological damage, a positive diagnosis of epilepsy, or having first-degree relatives diagnosed with epilepsy.
* Presence of a cardiac pacemaker or other metallic devices.
* Infectious or gastrointestinal disorders.
* Open facial wounds, motor or visual impairments, or neuromuscular pain that would prevent using the Oculus VR headset.
* Refusal to consent, either by the individual or their legal representative, for study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Feasibility based on the health staff operator perspective using the System Usability Scale (SUS) | From enrollment to the end of treatment at 3 weeks
  The SUS scale permitted the obtaining of information about the system's usability. The SUS range raw score from 0 to 100.
Feasibility using an Ad-hoc questionnaire | From enrollment to the end of treatment at 3 weeks
  The ad-hoc questionnaire permitted information about usability, engagement, satisfaction, and pleasure during exposure to the VR environment, as well as feelings and relaxation. The questionnaire is composed of 30 items based on a Likert scale from 1 to 5 (range score from 0 to 4), 15 items based on a Likert scale from 1 to 4 (range score from 0 to 3), and five open-ended questions.
Feasibility using the Non-pharmacological Therapy Experience Scale (NPT-ES) | From enrollment to the end of treatment at 3 weeks
  The NPT-ES permitted obtaining information about the subjective experience during the administration of non-pharmacological therapy. Five items are assessed on a Likert scale from 0 to 3. The total raw score is from 0 to 15.
Feasibility based on the health staff operator perspective using Focus Groups | From enrollment to the end of treatment at 3 weeks

SECONDARY OUTCOMES:
Assessment of the Responsive Behaviors administering the COHEN MANSFIELD - AGITATION INVENTORY (CMAI) | From enrollment to the end of treatment at 3 weeks
  The CMAI was permitted to obtain information about the frequencies of 29 different responsive behaviors based on a Likert scale from 0 to 6. The total raw score is from 0 to 174.
Assessment of the Responsive Behaviors administering the Functional Assessment Staging Tool (FAST) | From enrollment to the end of treatment at 3 weeks
  The FAST is a scale that permits the definition of the severity of functional impairment related to a diagnosis of cognitive impairment. It comprises seven degrees of severity and is assessed by the clinical health staff based on the anamnestic information.
Investigation of Adverse Symptoms Associated with Exposure to the Virtual Reality Device using the Virtual Reality Symptoms Questionnaire (VRSQ) | From enrollment to the end of treatment at 3 weeks
  The VRSQ assesses the general and eye-related physical symptoms of exposure to a virtual reality environment. The score assigned to each item ranges from 0 to 6, with a maximum total score of 84 (48 for general symptoms and 36 for eye symptoms). Higher scores represent worse symptoms, with 0 corresponding to no adverse effects and 84 to serious adverse effects.
Pain experience assessment using the Pain Assessment in Advanced Dementia (PAINAD) | From enrollment to the end of treatment at 3 weeks
  The PAINAD provides a method of analyzing the pain experienced by people with dementia. The total score ranges from 0-10 points.
Assessment of the pharmacotherapy administration and the users'behaviors before or during the VR sessions using the DataSheet 2 | From enrollment to the end of treatment at 3 weeks
  DataSheet 2 permits obtaining information about the administration of pharmacotherapy before, during, or after the VR exposure based on three open-ended questions filled out by the health staff operator that administers the experimental procedure. Moreover, the scale permitted information about the user's behavior during the VR exposure to be assessed by the health staff operator based on five questions on a Likert scale from 0 to 3 (Total raw score from 0 to 15).
Assessment of the state-anxiety using the State-Trait Anxiety Inventory-Y1 (STAI-Y1) | From enrollment to the end of treatment at 3 weeks
  The modified version of the (STAI-Y1), inspired by Appel et al.2021, was administered in this study to obtain information on the state-anxiety level and other types of emotions individuals experienced before and after the VR session. The current study will investigate relaxation, worry/anxiety, sadness, tightness, annoyance, and anger explicitly. The scale is administered as an interview based on a 5-point Likert scale from 1 (not at all) to 5 (a lot).
Emotional and behavioral assessment using the Observed Emotion Rating Scale (OERS) | From enrollment to the end of treatment at 3 weeks
  The OERS assess the presence and frequency of negative emotions (fear, anxiety, anger, and sadness) and positive (pleasure) feelings experienced during the session based on a scale from 1 to 5 (1: "undetected emotion"; 2: "emotion observed for less than 16 s"; 3: "emotion observed for 16-59 s"; 4: "emotion observed for 1-5 min"; 5: "emotion observed for more than 5 min").

OTHER OUTCOMES:
Assessment of Socio-demographic features using the Socio-demographic sheet | From enrollment to the end of treatment at 3 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- APSP ''Grazioli'', Trento, Italy, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pardini S, Gios L, Dianti M, Genovese A, Lamon M, Marcon J, Forti S, Mayora-Ibarra O. Exploring customised virtual environments in patients with cognitive decline and responsive behaviours: protocol for a proof-of-concept and feasibility study in a long-term care facility (iEMBRACE). BMJ Open. 2025 Dec 5;15(12):e098051. doi: 10.1136/bmjopen-2024-098051. PMID 41360455